CLINICAL TRIAL: NCT00638456
Title: Use of Topical Budesonide in the Treatment of Eosinophilic Esophagitis, a Randomized Clinical Trial
Brief Title: Use of Topical Budesonide in the Treatment of Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ranjan Dohil (Other)
Collaborators: Meritage Pharma, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ranjan Dohil, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VPI-106-01
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophils; Esophagitis; Microscopy
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis | interventions — Budesonide; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): oral viscous budesonide plus Prevacid
  Interventions: Drug: Budesonide plus Prevacid
- 2 (Placebo Comparator): placebo plus Prevacid
  Interventions: Drug: placebo plus Prevacid

INTERVENTIONS:
Drug: Budesonide plus Prevacid — Budesonide is taken daily for three months. In addition, Prevacid is taken twice daily for three months.
  Arms: 1
Drug: placebo plus Prevacid — Placebo is taken daily for three months. In addition, Prevacid is taken twice daily for three months.
  Arms: 2

SUMMARY:
This study is designed to evaluate whether or not oral viscous budesonide is effective in treating children with Eosinophilic Esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Histologic evidence of EE defined as greater than 20 eosinophils per hpf on esophageal biopsy
* Ages 1 yrs and older
* Ability to continue the same diet that the patient was on at the time of EGD with biopsy

Exclusion Criteria:

* Adverse reaction or allergy to budesonide
* Pregnancy
* Chronic diseases requiring immunomodulatory therapy
* Use of swallowed topical corticosteroids for EE within the past 3 months
* Use of systemic steroids 2 months prior to study entry
* Upper gastrointestinal bleed within 4 months of study entry
* Chronic use of medications that predispose to upper gastrointestinal bleeding including non-steroidal anti-inflammatory medications or anticoagulants
* Evidence of adrenal suppression prior to study entry
* Evidence of concurrent eosinophilic gastritis, enteritis, colitis, or proctitis
* Recent changes in asthma or allergic rhinitis therapy for 3 months

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjan Dohil, MD, Principal Investigator — UCSD
Locations (1):
- Rady Children's Hospital, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Dohil R, Newbury R, Fox L, Bastian J, Aceves S. Oral viscous budesonide is effective in children with eosinophilic esophagitis in a randomized, placebo-controlled trial. Gastroenterology. 2010 Aug;139(2):418-29. doi: 10.1053/j.gastro.2010.05.001. Epub 2010 May 7. PMID 20457157

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Viscous Budesonide Plus Prevacid: Budesonide plus Prevacid: Budesonide is taken daily for three months. In addition, Prevacid is taken twice daily for three months.
Period: Overall Study
Arm/Group | Oral Viscous Budesonide Plus Prevacid | Placebo Plus Prevacid
Started | 21 | 11
Completed | 15 | 9
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Viscous Budesonide Plus Prevacid | Placebo Plus Prevacid | Total
Number analyzed (Participants) | 21 | 11 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 11 | 32
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 17 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement of Espohageal Eosinophilia
Description: Repeat endoscopy was undertaken using the Olympus P160 endoscope (by RD) at 3 months of treatment.
Time Frame: 3 Months
Population: 6 subjects withdrew from the oral viscous budesonide plus Prevacid group and 2 withdrew from the placebo plus Prevacid group, and so they were not included in the data analsyis.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Viscous Budesonide Plus Prevacid | Placebo Plus Prevacid
Number analyzed (Participants) | 15 | 9
Participants | 13 | 0

2. Secondary Outcome: Upper Gastrointestinal Endoscopy Score
Description: Endoscopy scoring tool took into account the following categories:
  Mucosal pallor/reduced vasculature Linear furrows/mucosal thickening White plaques Concentric rings/stricture Friability/"tissue-paper" mucosa Histology scoring tools Epithelial histology score Peak eosinophil count
  Each category could score 0-3 for a total maximum score of 15. The higher the score the worse the disease.
Time Frame: Baseline and 3 Months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Oral Viscous Budesonide Plus Prevacid | Placebo Plus Prevacid
Number analyzed (Participants) | 15 | 9
units on a scale
  Baseline | 4.6 [0 to 9] | 7.8 [4 to 9]
  3 months | 1.5 [0 to 7] | 5.4 [1 to 9]

3. Secondary Outcome: Symptom Score
Description: Total score was based on the following symptoms:
  Heartburn/regurgitation Abdominal pain Nausea/vomiting Anorexia/early satiety Dysphagia Symptom induced nocturnal wakening Gastrointestinal bleeding
  Each symptom could score 0-2 for a maximum score for 14 points. The lower the score the milder the symptoms and the higher the score the more severe symptoms.
Time Frame: Baseline and 3 Months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Oral Viscous Budesonide Plus Prevacid | Placebo Plus Prevacid
Number analyzed (Participants) | 15 | 9
units on a scale
  Baseline | 3.5 [0 to 10] | 2.7 [1 to 6]
  3 months | 1.2 [0 to 7] | 1.8 [0 to 7]

ADVERSE EVENTS:
Arm/Group | Oral Viscous Budesonide Plus Prevacid | Placebo Plus Prevacid
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/11
Other Adverse Events (participants affected / at risk) | 3/21 | 5/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Viscous Budesonide Plus Prevacid (N=21) | Placebo Plus Prevacid (N=11)
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral Candida (Gastrointestinal disorders) | 1 (1) | 0 (0)
Trasient headache (Nervous system disorders) | 1 (1) | 1 (1)
Worsening Eczema (General disorders) | 0 (0) | 1 (1)
Chest Infection (Infections and infestations) | 0 (0) | 1 (1)
Mild Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
transient diarrehea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes